CLINICAL TRIAL: NCT03092232
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of Single Escalating Oral Doses Of Pf-06865571 In Healthy Adult Subjects
Brief Title: Single Dose Study to Assess the Safety, Tolerability and Pharmacokinetics(PK) of PF-06865571
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C2541001
Record Dates: First submitted 2017-03-02; First posted 2017-03-27 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Healthy
MeSH Terms: interventions — ervogastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1_Active and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo
- Cohort 2_Active and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo
- Cohort 3_Active and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo

INTERVENTIONS:
Drug: PF-06865571 — Single ascending dose of PF-06865571 as extemporaneously prepared solution/suspension, once every 2 week in a cross over study: 5 mg, 50 mg, 500 mg, TBD (to be determined)/2000 mg.
  Arms: Cohort 1_Active and Matching Placebo
Drug: PF-06865571 — Single ascending dose of PF-06865571 as extemporaneously prepared solution/suspension, once every 2 week in a cross over study: 15 mg, 150 mg, 1000 mg, TBD/2000 mg.
  Arms: Cohort 2_Active and Matching Placebo
Drug: PF-06865571 — Single repeated (TBD mg) dose as extemporaneously prepared solution/suspension of PF-06865571.
  Arms: Cohort 3_Active and Matching Placebo
Drug: Placebo — Matching Placebo for PF-06865571 for each cohort.

SUMMARY:
The current study is the first clinical trial proposed with PF-06865571. It is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) following administration of single doses of PF-06865571 to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and female of non-childbearing potential;
* Age of 18-55, inclusive;
* Body Mass Index 22.5 to 35.4 kg/m2, inclusive;
* Body weight >50 kg;
* Not on any prescription or non-prescription drugs within 7 days or 5 half-lives prior to first dose.

Exclusion Criteria:

* Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergises, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug test.
* History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary: (1)Aspartate aminotransferase (AST), alanine aminotransferase (ALT) level, or total bilirubin > upper limit of normal (ULN); (2) For optional Cohort 3 only, AST or ALT greater or equal to 1.5 × ULN, provided that data from Cohorts 1 and 2 support this limit; (3) • Subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is less than or equal to ULN plus ALT and AST are less than or equal to ULN plus alkaline phosphatase, hemoglobin, and reticulocyte count are all less than or equal to ULN.
* Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
* Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | Screening up to 35 days after last dose of study medication
  Number of participants with reported adverse events
Number of subjects with laboratory tests findings of potential clinical importance | Baseline (Day 0) up to 14 days after last dose of study medication
  Number of participants with potentially clinically important laboratory test findings
Number of subjects with vital signs findings of potential clinical importance | Baseline (Day 0) up to 14 days after last dose of study medication
  Number of participants with potentially clinically important vital sign measurements
Number of subjects with electrocardiogram (ECG) findings of potential clinical importance | Baseline (Day 0) up to 14 days after last dose of study medication
  Number of participants with potentially clinically important ECG findings

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  AUC (0-infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Dose normalized AUClast for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  dose normalized AUC will be analysed using a mixed model appropriate to the study design
Dose normalized AUCinf for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  Following log-transformation, dose normalized AUCinf will be analysed using a mixed model appropriate to the study design.
Maximum Observed Plasma Concentration (Cmax) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  Maximum Observed Plasma Concentration (Cmax)
Dose normalized Cmax for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  Following log-transformation, dose normalized Cmax will be analysed using a mixed model appropriate to the study design.
Time to Reach Maximum Observed Concentration for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  Plasma Decay Half-Life (t1/2)
Apparent Oral Clearance (CL/F) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post dose in each period
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C2541001&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+To+Assess+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Single+Escalating+Oral+Doses+Of+Pf-06865571+In+Healthy+Adult+Subjects